CLINICAL TRIAL: NCT00435591
Title: A Phase 4, Randomized, Parallel Group, Multi-Center Study to Assess the Safety and Efficacy of Multiple Dosing Regimens of IV Conivaptan in Subjects With Euvolemic or Hypervolemic Hyponatremia
Brief Title: A Study of Multiple Dosing Regimens of IV Conivaptan in Subjects With Euvolemic or Hypervolemic Hyponatremia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cumberland Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 087-CL-084
Record Dates: First submitted 2007-02-14; First posted 2007-02-15 (Estimated); Results first posted 2010-05-26 (Estimated); Last update posted 2014-05-15 (Estimated); Status verified 2014-04

CONDITIONS: Hyponatremia; Euvolemia; Hypervolemia
Keywords: Hyponatremia; Euvolemia; Hypervolemia; Conivaptan; Vaprisol®; YM087
MeSH Terms: conditions — Hyponatremia; Edema | interventions — conivaptan

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Dose Regimen 1 (Experimental): Placebo loading dose + 20mg/day continuous infusion conivaptan per ampoule
  Interventions: Drug: Conivaptan; Drug: placebo
- Dose Regimen 2 (Experimental): Conivaptan loading dose (20mg)+ 20mg/day continuous infusion conivaptan per ampoule
  Interventions: Drug: Conivaptan
- Dose Regimen 3 (Experimental): Placebo loading dose + 20mg/day continuous infusion conivaptan per premix bag
  Interventions: Drug: Conivaptan; Drug: placebo
- Dose Regimen 4 (Experimental): Conivaptan loading dose (20mg) + 20mg/day continuous infusion conivaptan per premix bag
  Interventions: Drug: Conivaptan

INTERVENTIONS:
Drug: Conivaptan — ampoule or premix bag
  Other Names: YM087; Vaprisol
Drug: placebo — ampoule or premix bag
  Arms: Dose Regimen 1; Dose Regimen 3

SUMMARY:
The study will evaluate the effectiveness and safety of multiple dosing regimens of IV conivaptan in subjects with euvolemic or hypervolemic hyponatremia

ELIGIBILITY:
Inclusion Criteria:

* Subject has a serum sodium value between 115 and 133 mEq/L
* Subject is euvolemic or hypervolemic

Exclusion Criteria:

* Clinical evidence of volume depletion or dehydration
* Uncontrolled brady- or tachyarrhythmias requiring emergent pacemaker placement or treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2007-01; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Art Wheeler, MD, Study Director — Cumberland Pharmaceuticals, Inc.
Locations (15):
- Charleston, South Carolina, United States
- India (4):
  - Bangalore
  - Bhopal
  - Hyderabaad
  - Karnāl
- Israel (10):
  - Afula
  - Ashkelon
  - Haifa
  - Holon
  - Jerusalem
  - Rehovot
  - Safed
  - Tel Aviv
  - Tel Litwinsky
  - Ẕerifin

REFERENCES:
- [Background] Kalra S, Efrati S, Arthur JM, Oliven A, Velez JC, McNutt BE, Klasen S, Abeyratne A. Effect of loading dose and formulation on safety and efficacy of conivaptan in treatment of euvolemic and hypervolemic hyponatremia. Am J Health Syst Pharm. 2011 Apr 1;68(7):590-8. doi: 10.2146/ajhp100243. PMID 21411800
- See also: Link to Prescribing Information — http://www.astellas.us/docs/vaprisol.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Dose Regimen 3: Placebo loading dose + 20 mg/day continuous infusion conivaptan per premix bag
- Dose Regimen 4: Conivaptan loading dose (20 mg) + 20 mg/day continuous infusion conivaptan per premix bag
Period: Overall Study
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4
Started | 30 | 31 | 30 | 30
Safety Analysis Set | 28 | 30 | 30 | 29
Full Analysis Set | 28 | 29 | 30 | 29
End of Treatment | 25 | 27 | 27 | 23
Completed | 23 | 27 | 25 | 19
Not Completed | 7 | 4 | 5 | 11

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4 | Total
Number analyzed (Participants) | 28 | 30 | 30 | 29 | 117
Age, Continuous [Mean (Standard Deviation); unit: years] — Population represented is Safety Analysis Set (SAF)
  years | 59.1 (20.28) | 61.1 (20.14) | 64.8 (14.13) | 63.3 (22.31) | 62.1 (19.28)
Sex: Female, Male [Count of Participants; unit: Participants] — Population represented is Safety Analysis Set (SAF)
  Participants
    Female | 14 | 13 | 16 | 18 | 61
    Male | 14 | 17 | 14 | 11 | 56
Race/Ethnicity, Customized [Number; unit: Participants] — Population represented is Safety Analysis Set (SAF)
  Participants
    White | 14 | 16 | 14 | 16 | 60
    Black/ African -American | 0 | 1 | 0 | 0 | 1
    Asian | 14 | 13 | 15 | 13 | 55
    American Indian / Alaskan | 0 | 0 | 1 | 0 | 1
Volume Status/ Underlying Cause of Hyponatremia [Number; unit: Participants] — Population represented is Safety Analysis Set (SAF)
  SIADH: Syndrome of inappropriate antidiuretic hormone secretion CHF: Congestive heart failure COPD: Chronic obstructive pulmonary disease
  Participants
    Euvolemic/ SIADH | 15 | 11 | 11 | 9 | 46
    Euvolemic/ CHF | 1 | 0 | 0 | 0 | 1
    Euvolemic/ Malignancy | 0 | 1 | 3 | 0 | 4
    Euvolemic/ Idiopathic | 0 | 1 | 1 | 2 | 4
    Euvolemic/ COPD | 1 | 0 | 0 | 0 | 1
    Euvolemic/ Unknown | 6 | 8 | 8 | 10 | 32
    Euvolemic/ Other | 2 | 7 | 4 | 6 | 19
    Hypervolemic/ SIADH | 0 | 0 | 1 | 0 | 1
    Hypervolemic/ CHF | 3 | 2 | 0 | 2 | 7
    Hypervolemic/ Unknown | 0 | 0 | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number and Severity of Infusion Site Reactions (ISRs) Using a Modified ISR Reporting Scale for Phlebitis and Infiltration in Patients Treated With Dose Regimen 1 and Dose Regimen 2
Description: Infusion Site Reaction (ISR) was any local event other than isolated pain, bleeding, or bruising at the site of infusion.
  One ISRMS has been reported for each participant & represents the most severe state of ISR for that participant.
  ISR scale is a health care provider assessment of ISRs using the following modified 5 point reporting scale: 0= No new reaction; 1+=Infusion site erythema, infusion site pain, infusion site warmth; 2+= Infusion site edema; 3+=Phlebitis, venous induration; 4+=Thrombophlebitis, venous thrombosis, infusion site infection, infusion site cellulitis
Time Frame: 48 hours
Population: Population is Safety Analysis Set (SAF): All randomized patients who received at least 1 dose of study drug.
  The number of participants per arm is consistent for all categories of the data table.
Measure: Number; unit: Participants
Arm/Group | Dose Regimen 1 | Dose Regimen 2
Number analyzed (Participants) | 28 | 30
Participants
  Infusion Site Reaction - No assessment | 0 | 1
  Infusion Site Reaction - 0 | 17 | 16
  Infusion Site Reaction - 1+ | 5 | 7
  Infusion Site Reaction - 2+ | 2 | 0
  Infusion Site Reaction - 3+ | 4 | 5
  Infusion Site Reaction - 4+ | 0 | 1
Statistical Analysis 1: Comparison: Dose Regimen 1 vs Dose Regimen 2; Aggregated data were used to determine differences between groups. Statistical analysis is relevant to the aggregated data of all rows except the "no assessment" row; Test type: Superiority or Other; Least Squares Mean Difference = 0.23, 95% CI 2-sided [-0.37 to 0.83]

2. Secondary Outcome: Change From Baseline in Serum Sodium at Each Time Point Over the Duration of the Treatment Period and 7-day Post Treatment Period
Description: Baseline serum sodium value is the average of 2 serum sodium values taken at least 4 hours apart on Day-1 and within 24 hours of Hour 0 in the Treatment Period.
  Change from Baseline is calculated as Time point minus Baseline.
Time Frame: Baseline at 4, 6, 10, 16, 24, 30, 40, 48.5 hours and 7 days post-treatment
Population: Population is Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study drug and who had both baseline and postbaseline serum sodium data.
  The number of participants analyzed per arm represents Full Analysis Set. The numbers of participants for each time point are noted in the category titles.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4
Number analyzed (Participants) | 28 | 29 | 30 | 29
mmol/L
  Baseline | 124.6 (3.75) | 123.5 (4.08) | 124.5 (3.67) | 124.0 (4.63)
  Change at Hour 4 (N=28; 26; 30; 28) | 1.2 (3.67) | 1.5 (2.67) | 0.7 (2.13) | 1.9 (3.92)
  Change at Hour 6 (N=27; 27; 29; 27) | 1.1 (1.96) | 2.5 (2.88) | 1.5 (2.70) | 2.7 (3.23)
  Change at Hour 10 (N=27; 28; 30; 26) | 2.3 (2.92) | 2.9 (3.09) | 2.7 (3.88) | 2.9 (3.40)
  Change at Hour 16 (N=24; 24; 27; 23) | 2.0 (2.93) | 4.0 (4.09) | 4.2 (3.82) | 4.8 (3.90)
  Change at Hour 24 (N= 27; 27; 30; 24) | 3.3 (3.23) | 4.5 (3.85) | 4.4 (4.43) | 5.0 (3.81)
  Change at Hour 30 (N=27; 28; 28; 23) | 3.1 (4.13) | 4.5 (3.51) | 4.8 (4.14) | 4.1 (2.81)
  Change at Hour 40 (N=24; 26; 26; 24) | 4.3 (3.01) | 5.1 (4.14) | 6.9 (4.68) | 6.1 (4.52)
  Change at Hour 48.5 (N=26; 28; 28; 27) | 4.6 (4.01) | 5.8 (4.63) | 6.5 (4.19) | 5.4 (4.37)
  Change at Day 7 (N=23; 27; 25; 17) | 6.7 (5.87) | 9.6 (5.17) | 7.2 (4.22) | 8.9 (5.11)

3. Secondary Outcome: Baseline Adjusted Area Under the Concentration - Time Curve (AUC) in Serum Sodium Over the Duration of the First 24.5 Hours, the First 48.5 Hours, and the First 96.5 Hours
Description: AUCna t is calculated as the baseline-adjusted area under serum sodium levels for a duration of time 0 to time t.
  Baseline serum sodium value is the average of 2 serum sodium values taken at least 4 hours apart on Day-1 and within 24 hours of Hour 0 in the Treatment Period.
Time Frame: 24.5 hours, 48.5 hours and 96.5 hours
Population: Population is Full Analysis Set (FAS): All randomized patients who received at least 1 dose of study drug and who had both baseline and postbaseline serum sodium data.
  The number of participants per arm is consistent for all categories of the data table.
Measure: Mean (Standard Deviation); unit: hr * mEq/L
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4
Number analyzed (Participants) | 28 | 29 | 30 | 29
hr * mEq/L
  AUCna at 24.5 hours | 45.600 (55.919) | 70.569 (73.042) | 66.096 (73.662) | 82.470 (82.195)
  AUCna at 48.5 hours | 133.664 (127.156) | 194.561 (166.015) | 205.522 (163.261) | 207.043 (170.153)
  AUCna at 96.5 hours | 375.379 (331.298) | 503.127 (340.247) | 558.926 (351.718) | 528.377 (371.075)

4. Secondary Outcome: Time From the First Dose of Study Drug to a Confirmed > 4 mEq/L Increase From Baseline in Serum Sodium During the 48.5 Hour Treatment Period
Description: The upper limits of the interquartile range were not estimable in three of the treatment arms. Only the "placebo loading dose + YM087 premix continuous infusion" arm will be reported.
  Time is number of hours to reach an increase of exceeding 4 mEq/L from baseline serum sodium.
  Baseline serum sodium value is the average of 2 serum sodium values taken at least 4 hours apart on Day-1 and within 24 hours of Hour 0 in the Treatment Period.
Time Frame: 48.5 hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Hours
Arm/Group | Dose Regimen 3
Number analyzed (Participants) | 30
Hours | 24.08 [16.00 to 40.50]

5. Secondary Outcome: Number of Patients With Confirmed Serum Sodium Level Exceeding 4 mEq/L Increase From Baseline Over the Duration 0-24.5 Hours, 0-48.5 Hours, and 0-96.5 Hours
Description: Patients with confirmed serum sodium level exceeding 4 mEq/L increase from baseline.
  Baseline serum sodium value is the average of 2 serum sodium values taken at least 4 hours apart on Day-1 and within 24 hours of Hour 0 in the Treatment Period.
Time Frame: 0-24.5 hours, 0-48.5 hours and 0-96.5 hours
Population: as for outcome 3
Measure: Number; unit: Participants
Groups:
- Dose Regimen 4: Conivaptan loading dose (20mg)+20mg/day continuous infusion conivaptan per premix bag
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4
Number analyzed (Participants) | 28 | 29 | 30 | 29
Participants
  0 - 24.5 Hours | 6 | 13 | 13 | 10
  0 - 48.5 Hours | 13 | 15 | 23 | 19
  0 - 96.5 Hours | 21 | 22 | 27 | 24

6. Secondary Outcome: Number of Patients With Confirmed Serum Sodium Level Exceeding 6 mEq/L Increase From Baseline or Confirmed Normal Serum Sodium Level Exceeding 135 mEq/L Over the Duration 0-24.5 Hours, 0-48.5 Hours, and 0-96.5 Hours
Description: Patients with confirmed serum sodium level exceeding 6 mEq/L increase from baseline or confirmed normal serum sodium level exceeding 135 mEq/L.
  Baseline serum sodium value is the average of 2 serum sodium values taken at least 4 hours apart on Day-1 and within 24 hours of Hour 0 in the Treatment Period.
Time Frame: 0-24.5 hours, 0-48.5 hours and 0-96.5 hours
Population: as for outcome 3
Measure: Number; unit: Participants
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4
Number analyzed (Participants) | 28 | 29 | 30 | 29
Participants
  0 - 24.5 Hours | 1 | 6 | 7 | 6
  0 - 48.5 Hours | 6 | 13 | 17 | 12
  0 - 96.5 Hours | 13 | 16 | 24 | 19

ADVERSE EVENTS:
Description: Numbers of Participants at Risk represent the Safety Analysis Set (SAF).
  AE collection began at the start of study drug infusion and continued through Post Treatment Period Day 7. AEs collected in this time interval were defined as treatment emergent AEs (TEAEs) for patients who completed or prematurely discontinued study drug.
Arm/Group | Dose Regimen 1 | Dose Regimen 2 | Dose Regimen 3 | Dose Regimen 4
Serious Adverse Events (participants affected / at risk) | 2/28 | 5/30 | 8/30 | 2/29
Other Adverse Events (participants affected / at risk) | 6/28 | 12/30 | 4/30 | 8/29
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Regimen 1 (N=28) | Dose Regimen 2 (N=30) | Dose Regimen 3 (N=30) | Dose Regimen 4 (N=29)
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0
Collapse of lung (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 0 | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Haemodialysis (Surgical and medical procedures) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Regimen 1 (N=28) | Dose Regimen 2 (N=30) | Dose Regimen 3 (N=30) | Dose Regimen 4 (N=29)
Anaemia (Blood and lymphatic system disorders) | 0 | 4 | 0 | 0
Constipation (Gastrointestinal disorders) | 3 | 5 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 6 | 0 | 4
Chest pain (General disorders) | 2 | 0 | 2 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 4
Headache (Nervous system disorders) | 3 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 2 | 0 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 2

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the currency or completeness of the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document. Sponsor may delay the publication for an additional 60 days to seek patent protection.